CLINICAL TRIAL: NCT04932356
Title: To Evaluate the Impact of a Telephone Therapeutic Education Program in DM2 Patients With Poor Metabolic Control Over Glycosylated Hemoglobin and Spontaneous Nursing Visits, in a Primary Care Center
Brief Title: Telephone Therapeutic Education Program in DM2 Patients With Poor Metabolic Control
Acronym: TTEDMV1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mª Dolores Rodríguez Garrido (Other)
Responsible Party: Sponsor-Investigator, Mª Dolores Rodríguez Garrido, Principal investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Organization: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4R16/146
Record Dates: First submitted 2021-06-12; First posted 2021-06-21 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Educational Technology; Diabetes Mellitus Type 2; Glycated Hemoglobin A; Pragmatic Clinical Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Fortnightly reinforcement of diabetes education, diet review, exercise, emotional support, doubts with insulin or oral medication and the registration of blood glucose controls, through telephone calls scheduled at a specific time during a semester.
Masking Description: Patients will be randomly assigned to each group at the beginning of recruitment. Patients who are in the intervention group will be aware of the group in which they are because it requires biweekly telephone visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Education by phone (Other): Therapeutic education in diabetes mellitus (pharmacological, nutritional, physical exercise, social adherence ... etc) on face-to-face visit and then reinforcement each 15 days over the weak points of this visit.
  Interventions: Other: Therapeutic education by phone
- Traditional Therapeutic Education (Other): Therapeutic education in diabetes mellitus (pharmacological, nutritional, physical exercise, social adherence ... etc) on face-to-face visit.
  Interventions: Other: Therapeutical education traditional

INTERVENTIONS:
Other: Therapeutic education by phone — The patients who participate in the intervention group, after their face-to-face visit, will undergo a fortnightly reinforcement by telephone of diabetes education (review of diet, physical exercise, doubts about insulin or oral medication and the registry of blood glucose controls). In addition, emotional support will be provided to the patient, along with a semester calendar with scheduled calls to carry out the intervention, at a specific time.
  Arms: Therapeutic Education by phone
Other: Therapeutical education traditional — The patients participating in the study will be visited in person every six months where the control group will follow the usual protocol of the health center in the face-to-face visits, with their respective analyzes and pertinent tests, together with health education and adherence to pharmacological treatment.
  Arms: Traditional Therapeutic Education

SUMMARY:
Diabetes Mellitus (DM) is one of the most prevalent chronic diseases worldwide and with a significant impact on health spending.

The literature identifies that the telephone improves the process of clinical care and patient outcomes. Programs are known to have demonstrated improvements in HbA1c outcome in DM2.

In the majority of patients their follow-up is carried out from primary care, where they occupy a third of the visits, it is a main reason for consultation.

The mobile phone is becoming an interesting tool for therapeutic education.

The objective: To decrease the HbA1c value by 10% in patients who have their HbA1c >9% and 0.5% in those who have an HbA1c value <9%-Reduce the number of spontaneous visits in nursing consultations.

Know the attitude and motivations of the patients participating in the study It will be a probabilistic randomized intervention study at the Mas Font Primary Care Center in Viladecans (Barcelona).

According to medical history as of December 31, 2020, there were 1554 patients diagnosed with DM2, 402 DM2 patients with poor control (HbA1c >8%) Patients who meet inclusion criteria will be contacted by telephone or at consultations and will be offered to participate and sign consent.

They are then automatically randomized to intervention or control group. Study participants will be visited in person every six months and both groups will follow the center's protocol in face-to-face visits, The intervention group will be reinforced with a fortnightly telephone visit.

DETAILED DESCRIPTION:
The study is of the probabilistic random intervention type, in a Primary Care center. The area where the study will be carried out: Population attached to ABS Mas Font over 18 years (18,431 people), in Viladecans (Barcelona). In the computerized medical history database, as of December 31, 2020, 1554 patients diagnosed with DM2 were found. By 2020 they had two HBa1cs registered in 402 patients (26% of all PATIENTS with DM2), only 711 (45.75%) 441 (28.4%) no. With one of the last two > 8 there are 145 patients. With the last two values > 8 there are 87 patients. Socio-economic data Typology according to CatSalut - Urban population with medium-high privacy MEDEA* ABS Viladecans Index 1 x 0'70 (Median of Catalonia 0'44) *It is a deprivation rate based on the following socio-economic indicators: manual workers, unemployment, eventual employees, total under-education and in 18 young people. Inclusion and exclusion criteria the denial of participating in the study. Sample calculation In the computerized medical history database, as of December 31, 2020, 1554 patients diagnosed with DM2 were consisting of 402 DM2 patients (26%) have at least two records of HbA1c. Accepting an alpha risk of 5%, beta less than 20%, in a unilateral contrast and waiting to detect a minimum difference of 0.9, for a deviation of 1.2 in HBa1c values and with losses not greater than 10%, 32 patients are required in each group. The sample should be increased by 20% in case there were drop outs, requiring a sample of 38 patients in each group to be able to find a difference in HbA1c. (IMIM GRANMO https://www.imim.es/ofertadeserveis/software-public/granmo/) Source of subjects From the list of patients who meet criteria you will get a sample Random. The collected patients will be contacted by telephone or at the consultations and offered to participate in the study. The purpose of the same will be explained and the confidentiality of the data will be ensured. If they agree to participate they will be summoned to the center where they sign the informed consent (see attached document). They are then automatically randomized to intervention or control group. Definition of variables Demographic:

-age: in Limitations and possible biases One limitation that we can find is that the data on the follow-up of the medication varies, since during a year the patient can change treatment, due to hospital admission (variable that will be collected in both groups and a stratified analysis will be performed if necessary).

The loss of follow-up of patients due to different causes (such as patients who can change cities during vacation periods and difficult telephone locations due to difficulties in coverage, changes of residence). The final impact of the study and the reason for the losses will be evaluated.

Lack of feedback between the patient and the nurse

ELIGIBILITY:
Inclusion Criteria:

* DM2 patient with HbA1c > of 8%
* With some form of drug medication for their diabetes.

Exclusion Criteria:

* persons with gestational diabetes,
* psychiatric disease
* hearing or vocalization problems,
* terminal patient in PADES,
* patient with chronic acute disease (MACA),
* the denial of participating in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c Result | 7 months
  Descriptive statistics of the variables will be carried out, using measures of central tendency and dispersion for quantitative variables and percentages with a 95% confidence interval for qualitative variables.
  A comparison of both groups will be carried out at the beginning of the study, using t-Student or chi-square according to the nature of the variables and if the application conditions allow it.
  Bivariate statistics will also be performed at the end of the study, to evaluate differences between both groups, and other independent variables, with respect to the outcome variables.
  Multivariate statistics will be performed, by means of logistic regression, using as the dependent variable having or not achieved the decrease in hemoglobin and as independent variables those that have shown significance at the bivariate level.

SECONDARY OUTCOMES:
patient motivation | 6 month
  To evaluate the motivation and attitude of the patient with respect to his diabetes, in the initial visit and at the end of the intervention, the DAS-3sp questionnaire will be used. The proposed motivations and attitudes test is validated by J.Mª Hernandez et al. 19 (annex two). Where the changes in the global score of the scale between the visit at the beginning and at the end of the intervention will be assessed, comparing the initial and final tests.

CONTACTS AND LOCATIONS:
Overall Officials: MªDolores Rodriguez, diploma, Principal Investigator — ICS
Locations (1):
- MªDolores Rodriguez, Viladecans, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] J.M. Hernández, J. Basora, X. Ansa, J.L. Piñol, M. Millan, D. Figuerola. La versión española de la Diabetes Attitude Scale (DAS-3sp): un instrumento de medición de actitudes y motivaciones en Diabetes. Endocrinol Nutr., 49 (2002), pp. 293-298
- [Background] Roca-Espino D, Orois-Añón A. El control de la diabetes a distancia. ¿Cuánto hay de verdaderamente útil bajo el término telemedicina? Avances en Diabetología 2015; 31(1):1-7.
- [Background] Picón César MJ. Documento de posicionamiento sobre el uso de la telemedicina aplicada a la atencion diabetologica. Avances en diabetología 2010;26(3):147-150.
- [Background] Zhou P, Xu L, Liu X, Huang J, Xu W, Chen W. Web-based telemedicine for management of type 2 diabetes through glucose uploads: a randomized controlled trial. Int J Clin Exp Pathol. 2014 Dec 1;7(12):8848-54. eCollection 2014. PMID 25674254
- [Result] Edmonds M, Bauer M, Osborn S, Lutfiyya H, Mahon J, Doig G, Grundy P, Gittens C, Molenkamp G, Fenlon D. Using the Vista 350 telephone to communicate the results of home monitoring of diabetes mellitus to a central database and to provide feedback. Int J Med Inform. 1998 Aug-Sep;51(2-3):117-25. doi: 10.1016/s1386-5056(98)00109-9. PMID 9794328
- [Result] Dennis SM, Harris M, Lloyd J, Powell Davies G, Faruqi N, Zwar N. Do people with existing chronic conditions benefit from telephone coaching? A rapid review. Aust Health Rev. 2013 Jun;37(3):381-8. doi: 10.1071/AH13005. PMID 23701944
- [Result] Kaur R, Kajal KS, Kaur A, Singh P. Telephonic Consultation and follow-up in Diabetics: Impact on Metabolic Profile, Quality of Life, and Patient Compliance. N Am J Med Sci. 2015 May;7(5):199-207. doi: 10.4103/1947-2714.157483. PMID 26110131
- [Result] Munshi MN, Segal AR, Suhl E, Ryan C, Sternthal A, Giusti J, Lee Y, Fitzgerald S, Staum E, Bonsignor P, DesRochers L, McCartney R, Weinger K. Assessment of barriers to improve diabetes management in older adults: a randomized controlled study. Diabetes Care. 2013 Mar;36(3):543-9. doi: 10.2337/dc12-1303. Epub 2012 Nov 27. PMID 23193208
- [Result] Izquierdo RE, Knudson PE, Meyer S, Kearns J, Ploutz-Snyder R, Weinstock RS. A comparison of diabetes education administered through telemedicine versus in person. Diabetes Care. 2003 Apr;26(4):1002-7. doi: 10.2337/diacare.26.4.1002. PMID 12663564
- [Result] Holtz B, Lauckner C. Diabetes management via mobile phones: a systematic review. Telemed J E Health. 2012 Apr;18(3):175-84. doi: 10.1089/tmj.2011.0119. Epub 2012 Feb 22. PMID 22356525
- [Result] Esmatjes E, Jansa M, Roca D, Perez-Ferre N, del Valle L, Martinez-Hervas S, Ruiz de Adana M, Linares F, Batanero R, Vazquez F, Gomis R, de Sola-Morales O; Telemed-Diabetes Group. The efficiency of telemedicine to optimize metabolic control in patients with type 1 diabetes mellitus: Telemed study. Diabetes Technol Ther. 2014 Jul;16(7):435-41. doi: 10.1089/dia.2013.0313. Epub 2014 Feb 14. PMID 24528195
- [Result] Klonoff DC. Using telemedicine to improve outcomes in diabetes--an emerging technology. J Diabetes Sci Technol. 2009 Jul 1;3(4):624-8. doi: 10.1177/193229680900300401. No abstract available. PMID 20144303
- [Result] Zolfaghari M, Mousavifar SA, Haghani H. Mobile phone text messaging and Telephone follow-up in type 2 diabetic patients for 3 months: a comparative study. J Diabetes Metab Disord. 2012 Aug 24;11(1):7. doi: 10.1186/2251-6581-11-7. PMID 23497735 (Retraction: PMID 23497527 J Diabetes Metab Disord. 2013 Mar 07;11(1):21)
- [Result] Zhai YK, Zhu WJ, Cai YL, Sun DX, Zhao J. Clinical- and cost-effectiveness of telemedicine in type 2 diabetes mellitus: a systematic review and meta-analysis. Medicine (Baltimore). 2014 Dec;93(28):e312. doi: 10.1097/MD.0000000000000312. PMID 25526482
- [Result] McGloin H, Timmins F, Coates V, Boore J. A case study approach to the examination of a telephone-based health coaching intervention in facilitating behaviour change for adults with Type 2 diabetes. J Clin Nurs. 2015 May;24(9-10):1246-57. doi: 10.1111/jocn.12692. Epub 2014 Oct 16. PMID 25319572
- [Result] Nuti L, Turkcan A, Lawley MA, Zhang L, Sands L, McComb S. The impact of interventions on appointment and clinical outcomes for individuals with diabetes: a systematic review. BMC Health Serv Res. 2015 Sep 2;15:355. doi: 10.1186/s12913-015-0938-5. PMID 26330299
- See also: Human Experimentation. Code of Ethics of the World Medical Association. Declaration of Helsinki. — http://www.ncbi.nlm.nih.gov/pubmed/14150898
- See also: Construcción de un índice de privación a partir de datos censales en grandes ciudades españolas: (Proyecto MEDEA). — https://scielo.isciii.es/pdf/gs/v22n3/original1.pdf
- See also: 10. Orozco-Beltrán D, et al. Abordaje de la adherencia en diabetes mellitus tipo 2: situación actual y propuesta de posibles soluciones. — http://dx.doi.org/10.1016/j.aprim.2015.09.001